CLINICAL TRIAL: NCT06244147
Title: Long Term Safety and Efficacy of KSM-66 Ashwagandha (Standardized Root Extract of Withania Somnifera) in Adults: A Prospective, Observational Study
Brief Title: Long Term Safety and Efficacy of KSM-66 Ashwagandha in Adults
Status: Completed | Type: Observational
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Other Study IDs: Ixoreal-Safety-CT-06-22
Record Dates: First submitted 2024-01-24; First posted 2024-02-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: All
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: KSM-66 Ashwagandha Root Extract — Participants will take KSM-66 Ashwagandha root extract 300mg twice a day for the duration of the study.

SUMMARY:
The primary objective is to evaluate the clinical safety of KSM-66 Ashwagandha (Withania Somnifera) on long-term administration over 12 months. The secondary objectives are to evaluate the laboratory safety of KSM-66 Ashwagandha (Withania Somnifera) on long-term administration over 12 months and to evaluate the efficacy of KSM-66 Ashwagandha (Withania Somnifera) on long-term administration over 12 months.

DETAILED DESCRIPTION:
To qualify for this study, participant must be male or female between 18 and 65 years old and prescribed KSM-66 Ashwagandha by their clinicians for a long-term period. Participants must have no plan to commence any other alternative treatment modality for their conditions. Participants must be willing to sign an informed consent document and to comply with all study related procedures. Participants must have a body mass index between 25 and 39.9 kg/m2.

In this study, a total of 200 subjects will be included across 4-5 study sites, for a total duration of 12 months. At the initial visit, prospective patients will be screened for enrollment based on the requirements of the study, medical history, and clinical examination. Before starting any study related procedures, participants will be explained about the study in detail and a written informed consent will be obtained from participants prior to participation in this study. This document is a part of the written informed consent procedure. A detailed medical history including the associated conditions will be recorded. A general and physical examination will be performed to detect any abnormal parameters. If participants meet the eligibility criteria, they will be enrolled in the study.

After enrollment in the study, participants will be asked to consume Ashwagandha 300 mg root extract capsule orally twice daily, morning and evening after breakfast and dinner with a glass of water. At Visit 1 (Screening/Enrollment/Baseline Visit - Day -3 to Day 0), demography and medical history will be taken, physical examination and vital signs will be performed, blood will be collected, study medication will be dispensed, and Clinical Global Impression - Improvement (CGI-I) scale and Quality of Life using the SF-12 QoL scale will be assessed.

At Visits 2 to 6 (Months 1, 2, 3, 4, 5), participants will follow up remotely via a phone call. Compliance and concomitant medication will be noted.

At Visit 7 (Month 7), participants will follow up on site, where a physical examination and vital signs will be performed, blood will be collected, study medication will be dispensed, Clinical Global Impression - Improvement (CGI-I) scale and Quality of Life using the SF-12 QoL scale will be assessed, and compliance will be assessed.

At Visits 8 to 12 (Months 7, 8, 9, 10, 11), participants will follow up remotely via a phone call. Compliance and concomitant medication will be noted.

At Visit 13 (Final Visit - Month 12), participants will follow up on site, where a physical examination and vital signs will be performed, blood will be collected, Clinical Global Impression - Improvement (CGI-I) scale and Quality of Life using the SF-12 QoL scale will be assessed, and compliance will be assessed. Participants will be monitored throughout the study, including any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male and female) aged between 18 and 65 years.
* Prescribed KSM-66 Ashwagandha by their clinicians for long-term period.
* No plan to commence any other alternative treatment modality for their conditions.
* Willingness to sign an informed consent document and to comply with all study related procedures.
* Participants with Body mass index between 25 and 39.9 kg/m2.

Exclusion Criteria:

* Patients receiving any of the medications known to affect stress and anxiety (corticosteroids, antidepressants, anti-psychotics, mood stabilizers, and anti-epileptic medications) during 4 weeks prior to screening.
* Patients currently (or within the past 4 weeks prior to screening) taking any over the counter use of herbal extracts such as Ginkgo Biloba, St. John's Wort, Omega-3 etc.
* Patients with depressive episode, suicidal tendency, panic disorder, social phobia, obsessive-compulsory disorder; alcohol dependency; schizophrenia and mania.
* Patients with known post-traumatic stress disorder (PTSD).
* Patients with known clinically significant acute unstable hepatic, renal, cardiovascular, or respiratory disease that will prevent participation in the study.
* Patients with known hypersensitivity to Ashwagandha.
* Patients who had participated in other clinical trials during previous 3 months.
* Patients who have any clinical condition, according to the investigator which does not allow safe fulfillment of clinical trial protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 subjects who are prescribed KSM-66 Ashwagandha by their clinicians for long-term period for their respective health conditions will be included for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Number and proportion of Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Event (TESAE) due to KSM-66 Ashwagandha (Withania Somnifera) over 12 months period

SECONDARY OUTCOMES:
Liver Parameters | 6 and 12 months
  Changes in laboratory values for serum alanine transaminase 6 months and 12 months after start of KSM-66 Ashwagandha
Liver Parameters | 6 and 12 months
  Changes in laboratory values for aspartate transaminase 6 months and 12 months after start of KSM-66 Ashwagandha
Liver Parameters | 6 and 12 months
  Changes in laboratory values for alkaline phosphatase 6 months and 12 months after start of KSM-66 Ashwagandha
Liver Parameters | 6 and 12 months
  Changes in laboratory values for bilirubin 6 months and 12 months after start of KSM-66 Ashwagandha
Renal Parameters | 6 and 12 months
  Changes in laboratory values for renal parameters (serum creatinine, blood urea nitrogen) 6 months and 12 months after start of KSM-66 Ashwagandha
Muscle Parameters | 6 and 12 months
  Changes in laboratory values for serum creatine phosphokinase-MB 6 months and 12 months after start of KSM-66 Ashwagandha
Sex Hormones | 6 and 12 months
  Changes in laboratory values for serum testosterone 6 months and 12 months after start of KSM-66 Ashwagandha
Muscle Parameters | 6 and 12 months
  Changes in laboratory values for muscle parameters (serum creatine phosphokinase-MB), thyroid parameters (serum TSH, T3 and T4), and sex hormones (serum testosterone) 6 months and 12 months after start of KSM-66 Ashwagandha
Thyroid Parameters | 6 and 12 months
  Changes in laboratory values for thyroid parameters (serum TSH, T3 and T4) 6 months and 12 months after start of KSM-66 Ashwagandha
Serum Cortisol and Testosterone | 6 and 12 months
  Changes in laboratory values for serum cortisol and serum testosterone 6 months and 12 months after start of KSM-66 Ashwagandha
Clinical Global Impression | 6 and 12 months
  Clinical Global Impression - Improvement scale (CGI-I) score 6 months and 12 months after start of KSM-66 Ashwagandha [The CGI-I scale measures the change in the patient's clinical status from a specific point in time using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change]
Quality of Life Score | 6 and 12 months
  Changes from baseline in the Quality of Life (SF-12 QoL) scores 6 months and 12 months after start of KSM-66 Ashwagandha

CONTACTS AND LOCATIONS:
Locations (1):
- SF Research Institute, San Francisco, California, United States

REFERENCES:
- [Derived] Salve J, Kale S, Prajapati BL, Sparavigna A, Savant M, Ademola J, Langade D. Safety of 12-Months Administration of Ashwagandha (Withania somnifera) Standardized Root Extract in Healthy Adults: A Prospective, Observational Study. Phytother Res. 2025 Oct 8. doi: 10.1002/ptr.70096. Online ahead of print. PMID 41063394